CLINICAL TRIAL: NCT00808392
Title: A Phase III, Observer-blind, Randomized, Controlled, Multicenter Study to Investigate Immunogenicity and Safety of Haemophilus Influenzae Type b Vaccine in 2 - 4 Months Old Healthy Infants in China, According to the Recommended Regimen of 3 Intramuscular Doses Given One Month Apart
Brief Title: Safety and Immunogenicity of a Monovalent Conjugated Vaccine Against Haemophilus Influenzae Type b
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: M37P2
Record Dates: First submitted 2008-12-12; First posted 2008-12-15 (Estimated); Last update posted 2011-12-29 (Estimated); Status verified 2011-12

CONDITIONS: Haemophilus Influenzae Type b
Keywords: vaccine; prevention; haemophilus influenzae type b; children
MeSH Terms: conditions — Haemophilus Infections

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- 1 (Experimental)
  Interventions: Biological: Haemophilus influenzae type b vaccine
- 2 (Active Comparator)
  Interventions: Biological: Commercial Haemophilus influenzae type b vaccine

INTERVENTIONS:
Biological: Haemophilus influenzae type b vaccine — 3 doses one month apart of Monovalent conjugated vaccine against Haemophilus influenzae type b vaccine
  Arms: 1
Biological: Commercial Haemophilus influenzae type b vaccine — 3 doses one month apart of Haemophilus influenzae type b vaccine.
  Arms: 2

SUMMARY:
This study will investigate safety and immunogenicity of a monovalent conjugated vaccine against Haemophilus influenzae type b in healthy children aged 2 to 4 months in China.

ELIGIBILITY:
Inclusion Criteria:

* Infants of either sex, aged 2 - 4 months
* In good health as determined by:

  * medical history
  * physical examination
  * clinical judgment of the investigator;
* Available for all visits scheduled in the study and able to comply with all study regulations
* For whom written informed consent has been obtained from at least one parent or legal guardian

Exclusion Criteria:

* Parent or legal guardian is unwilling or unable to give written informed consent to participate in study
* Infants who have received any other Haemophilus influenzae type b immunization dose before
* Infants who presented a previous disease potentially related to Haemophilus influenzae type b
* Infants who had household contact and/or intimate exposure in the previous 30 days to an individual with ascertained Haemophilus influenzae type b disease
* Premature (before 37th week of gestation) or birth weight less than 2500 g
* History of anaphylactic shock, asthma, urticaria or other allergic reaction after previous vaccinations or hypersensitivity to any vaccine component
* Fever ≥ 38.0 °C (axillary body temperature) or/and significant acute or chronic infection requiring systemic antibiotic or antiviral therapy within the past 7 days before enrollment
* Subjects with any serious chronic disease such as cardiac, neurological, metabolic, hematologic, or neoplastic disease
* Known/suspected immunodeficiency, or autoimmune disease, or any immunologic disorder
* Subjects with any neurological disorder, e.g., epilepsy or history of seizure disorder
* Subjects with a clinically significant genetic anomaly
* Treatment with corticosteroids or other immunosuppressive drugs
* Any previous treatment with parenteral immunoglobulin preparation, blood products, and/or plasma derivatives
* Any vaccination administered within one week (7 days) before enrollment and/ or any planned administration of any vaccine outside the Chinese routine vaccination program.
* Participation in any other investigational trial simultaneously
* Planned surgery during the study period
* Any condition, which, in the opinion of the investigator, might interfere with the evaluation of the study objective

Ages: 2 Months to 4 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 916 (Actual)
Dates: Start 2008-11; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Immunogenic response measured by detection of anti-PRP antibodies by IgG enzyme linked immunosorbent assay (ELISA). | 90 days

SECONDARY OUTCOMES:
Rates of local and systemic reactions, adverse events (AEs), and serious adverse events (SAEs) after each single vaccination dose will be evaluated. | 90 days

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - the CDC of Dingxing county(site no 02), Dingxing, Hebei
  - The CDC of Zhengding county(site no 01), Zhengding, Hebei